CLINICAL TRIAL: NCT01972880
Title: ASP1941 Pharmacokinetic Study - Verification of Bioequivalence Between ASP1941 New Tablets and ASP1941 Conventional Tablets -
Brief Title: A Study to Compare the Oral Absorption of ASP1941 Among Two Types of Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-7001
Record Dates: First submitted 2013-10-16; First posted 2013-10-31 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy; Plasma Concentration of ASP1941
Keywords: Open-label design; Bioequivalence; ASP1941
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tablet-1 (Experimental)
  Interventions: Drug: ASP1941
- tablet-2 (Active Comparator)
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — Oral
  Other Names: ipragliflozin

SUMMARY:
To assess the bioequivalence of a single dose of ASP1941 between tablet-1 and tablet-2 in a two-way crossover method in non-elderly healthy male subjects. In addition, the safety of these products will be assessed.

DETAILED DESCRIPTION:
This study is a open-label randomized two-way crossover study. A single dose of two types of ASP1941 tablets are given to non-elderly healthy male subjects (16 subjects for each group, 32 subjects in total).

In case the bioequivalence of the 2 formulations cannot be proved in this study due to insufficient number of subjects, an add-on subject study will be conducted in this clinical trial as needed. Same design and methodology are to be applied to this study and the add-on subject study. The add-on subject study may not be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Body weight (at screening) >=50.0 kg and < 80kg
* BMI >= 17.6 and < 26.4 (BMI = Weight (kg)/(Height (m))2)
* Healthy, as judged by the investigator/sub-investigator based on physical examinations (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital of the period 1 admission to immediately before study drug administration

Exclusion Criteria:

* Received or scheduled to receive any investigational drugs in other clinical trials or post-marketing studies within 120 days before the screening or during the period from screening to hospital admission of the period 1 (Day -1).
* Donated or scheduled to donate more than 400 mL of whole blood within 90 days before the screening, more than 200 mL of whole blood within 30 days before screening, blood components within 14 days before screening, or whole blood or blood components during the period from screening to hospital admission of the period 1 (Day -1).
* Received or scheduled to receive medications (including OTC drugs) within 7 days before hospital admission of the period 1 (Day -1).
* A deviation from the normal range of blood pressure, pulse rate, body temperature, or standard 12-lead ECG at screening or hospital admission of the period 1 (Day -1)
* Concurrent or previous drug allergies
* Development of upper gastrointestinal disease (e.g., nausea, vomiting, and stomachache) within 7 days before hospital admission of the period1 (Day-1)
* Concurrent or previous hepatic disease (e.g., viral hepatitis, drug-induced hepatic disorder, and hepatic function disorder)
* Concurrent or previous heart disease (e.g., congestive cardiac failure, angina pectoris, and arrhythmia requiring treatment)
* Concurrent or previous gastrointestinal disease (e.g., peptic ulcer and reflux esophagitis), except for a history of appendicitis
* Concurrent or previous renal disease (e.g., acute renal failure, glomerulonephritis, and interstitial nephritis), except for a history of renal calculus
* Concurrent or previous endocrine disease (e.g., hyperthyroidism and blood abnormal growth hormone)
* Concurrent or previous cerebrovascular disorder (e.g., cerebral infarction)
* Concurrent or previous severe ketosis, diabetic coma, or precoma
* Previous use of ASP1941

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of unchanged ASP1941 | Before study drug administration on the administration day (Day 1), and 0.25，0.5，1，1.5，2，2.5，3，4，5，6，8，10，12，24，36，48，72 hours after administration

SECONDARY OUTCOMES:
Safety assessed by vital signs (sitting blood pressure, sitting pulse rate, axillary body temperature), AEs (including subjective symptoms and objective findings), Laboratory tests (hematology, biochemistry, urinalysis) and 12-lead ECGs | Up to 5 days after each administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan